CLINICAL TRIAL: NCT02942108
Title: Piezoelectric Vibrations and Tissue, Cellular and Molecular Mechanisms of Oral Wound Healing After Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Bozidar Brkovic, DDS, MSc, PhD, Professor, DDS, PhD, Associate Professor, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36/20
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Tooth, Impacted
Keywords: piezolectric surgery; conventional surgery; lower third molars
MeSH Terms: conditions — Tooth, Impacted | interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- healthy, conventional surgery (Active Comparator): Surgical bone removal by conventional rotary burs in healthy patients during third molar surgery
  Interventions: Procedure: conventional surgery
- healthy, piezo surgery (Experimental): Surgical bone removal by piezoelectric vibrations in healthy patients during third molar surgery
  Interventions: Procedure: piezo surgery

INTERVENTIONS:
Procedure: piezo surgery
  Arms: healthy, piezo surgery
Procedure: conventional surgery
  Arms: healthy, conventional surgery

SUMMARY:
The aim of this clinical trial is to investigate and compare the effect of piezoelectric surgery on tissue, cellular and molecular level of oral surgical wound healing and postoperative outcomes (pain, swelling, trismus) after lower third molar surgery in healthy patients

ELIGIBILITY:
Inclusion Criteria:

* bilaterally symmetrically impacted lower third molars

Exclusion Criteria:

* presence of intraoral infection
* chronic orofacial pain
* pregnancy/ lactation
* heavy tobacco smokers
* alcohol/ drug abuse
* allergic reaction to medicaments used

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
SOD activity in alveolar bone specimen | immediately after surgery
  Activity of enzyme superoxide dismutase in bone specimens obtained during lower third molar surgery
VEGF levels in alveolar bone specimen | immediately after surgery
MMP-9 level in alveolar bone specimen | immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bozidar M Brkovic, DDS,PhD, Principal Investigator — School of Dental Medicine, University of Belgrade; Milan V Vucetic, PhD student, Principal Investigator — School of Dental Medicine, University of Belgrade; Marija S Milic, DDS, PhD, Principal Investigator — School of Dental Medicine, University of Belgrade
Locations (1):
- School of Dental Medicine, University of Belgrade, Belgrade, Serbia

REFERENCES:
- [Derived] Bailey E, Kashbour W, Shah N, Worthington HV, Renton TF, Coulthard P. Surgical techniques for the removal of mandibular wisdom teeth. Cochrane Database Syst Rev. 2020 Jul 26;7(7):CD004345. doi: 10.1002/14651858.CD004345.pub3. PMID 32712962